CLINICAL TRIAL: NCT01898793
Title: A Phase 1/2 Study of Cytokine-Induced Memory-Like NK Cells in Patients With AML or MDS
Brief Title: Cytokine-induced Memory-like NK Cells in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Society of Clinical Oncology (Other); American Society of Hematology (Other); Gabrielle's Angel Foundation (Other); The Leukemia and Lymphoma Society (Other); National Cancer Institute (NCI) (NIH); ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201401085; 5F32CA200253-02 (NIH)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Leukapheresis; Interleukin-2; aldesleukin; Interleukins; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells (Experimental): * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors over 5 hours on day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion over 15-60 minutes on day 0.
  * Interleukin-2: Patients receive aldesleukin SC every other day for 2 weeks starting on day 1 (total of 7 doses)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Biological: IL-2; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells (Experimental): * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors over 5 hours on day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion over 15-60 minutes on day 0.
  * Interleukin-2: Patients receive aldesleukin SC every other day for 2 weeks starting on day 1 (total of 7 doses)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Biological: IL-2; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Phase I Dose Level 3: Maximum NK cell/number kg (Experimental): * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors over 5 hours on day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion over 15-60 minutes on day 0.
  * Interleukin-2: Patients receive aldesleukin SC every other day for 2 weeks starting on day 1 (total of 7 doses)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Biological: IL-2; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Phase II (IL-2): Maximum NK cell/number kg (Experimental): The recipient will begin a lymphodepleting preparative regimen of fludarabine and cyclophosphamide on Day -6. The haploidentical donor identified by HLA matching of the immediate family members will undergo non-mobilized large volume (20-L) leukapheresis on Day -1, and the NK cell product will be infused into the recipient on Day 0. Subcutaneous IL-2 will begin approximately 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Biological: IL-2; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg (Experimental): * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors on Day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion on Day 0.
  * Subcutaneous ALT-803 will begin approximately 4 hours after the infusion and will continue for a total of 2 doses (Days 0 and 5).
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Drug: ALT-803; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Pediatric Cohort: Maximum NK cell/number kg (Experimental): * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors on Day -1
  * CIML NK Cells: Patients undergo CIML NK cell infusion on Day 0
  * Subcutaneous IL-2 will begin approximately 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Cytokine-induced killer cells; Biological: IL-2; Procedure: Peripheral blood for correlative studies; Procedure: Bone marrow for correlative studies
- Donors (No Intervention): -The haploidentical donor identified by HLA matching of the immediate family members (parents, siblings, and children) will undergo non-mobilized leukapheresis on Day -1. Peripheral blood mononuclear cells (PBMCs) will be collected using standard collection techniques.

INTERVENTIONS:
Drug: Fludarabine
  Other Names: 2-F-ara-AMP; 75607-67-9; 9H-purin-6-amine; 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl); Beneflur; Fludara; fludarabine-5'-monophosphate
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Drug: Cyclophosphamide
  Other Names: Cytoxan®; CPM
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Procedure: Leukapheresis
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Biological: Cytokine-induced killer cells
  Other Names: CIK cells
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Biological: IL-2
  Other Names: Proleukin; recombinant human interleukin-2; recombinant interleukin-2; Ro-236019; T-cell growth factor; TCGF; TCGF,; interleukin; Aldesleukin
  Arms: Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Drug: ALT-803
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg
Procedure: Peripheral blood for correlative studies — -Screening, Day 0 prior to CIML NK infusion, Day 1, Day 3, Day 7, Day 8, Day 10, Day 14, Day 21, Day 28, Day 42, Day 60, Day 100, 6 months, 9 months, 12 months, and at disease relapse
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg
Procedure: Bone marrow for correlative studies — -Screening, Day 8, Day 14, Day 28, Between Day 42 and 60, Day 100, at disease relapse
  Arms: Lead-in Cohort & Phase II (ALT-803): Maximum NK cell/number kg; Pediatric Cohort: Maximum NK cell/number kg; Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK cells; Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK cells; Phase I Dose Level 3: Maximum NK cell/number kg; Phase II (IL-2): Maximum NK cell/number kg

SUMMARY:
This phase I/2 trial studies the side effects and best dose of activated natural killer cells in treating patients with relapsed or refractory acute myeloid leukemia and myelodysplastic syndromes. Giving chemotherapy before a donor natural killer cell infusion helps stop the growth of cancer cells and stops the patient's immune system from rejecting the donor's natural killer cells. Modified natural killer cells may help the body build an immune response to kill cancer cells. Aldesleukin (interleukin-2) may stimulate the white blood cells (including natural killer cells) to kill leukemia cells.

In the phase II and pediatric portion of the study, the investigators intend to use maximal tolerated or tested (MT/TD) CIML NK cell dose as determined from the phase I part of this study. The phase II portion of the study also replaces IL-2 with ALT-803. The rationale for this change is to support the donor derived NK cells in vivo after adoptive transfer.

With amendment 16, the decision was made to return to the use of rhIL-2 support instead of ALT-803.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis requirement for phase I patients:

  * Refractory AML without complete remission (CR) after induction therapy (primary induction failure) or relapsed AML after obtaining a CR.
  * OR High-risk AML (by ELN criteria; See Appendix C) in complete remission (CR) and has either refused hematopoietic stem cell transplantation OR is currently not eligible for hematopoietic stem cell transplantation OR for whom hematopoietic stem cell transplantation is being reserved for later relapse. This is inclusive of patients with minimal residual disease evidenced by cytogenetics, molecular testing, and/or flow cytometry.
  * OR Myelodysplastic syndrome (MDS) with excess blasts (>5%) and progressive disease at any time after initiation of DNA hypomethylator treatment during the past 2 years, OR failure to achieve complete or partial response or hematological improvement (see section 12.4) after at least six cycles of azacytidine or four cycles of decitabine administered during the past 2 years, OR intolerance to azacytidine or decitabine. MDS patients with isolated 5q- abnormalities that meet these criteria after lenalidomide therapy and DNA hypomethylator therapy are also eligible.
* Diagnosis requirement for phase II patients:

  *Refractory AML without CR after induction therapy (primary induction failure) or relapsed AML after obtaining a CR. Favorable-risk core binding factor (CBF) mutated AML and acute promyelocytic leukemia (APL) will be excluded.
* Diagnosis requirement for pediatric cohort patients:

  *Refractory AML without complete remission (CR) after induction therapy (primary induction failure) or relapsed AML after obtaining a CR.
* Age requirement for phase I and phase II patients: At least 18 years of age.
* Age requirement for pediatric cohort: 2-17 years of age.
* Available HLA-haploidentical donor that meets the following criteria:

  * Related donor (parent, sibling, offspring, or offspring of sibling)
  * At least 18 years of age
  * HLA-haploidentical donor/recipient match by at least Class I serologic typing at the A&B locus.
  * In general good health, and medically able to tolerate leukapheresis required for harvesting the NK cells for this study.
  * Negative for hepatitis, HTLV, and HIV on donor viral screen
  * Not pregnant
  * Voluntary written consent to participate in this study
* Patients with known CNS involvement with AML are eligible provided that they have been treated and CSF is clear for at least 2 weeks prior to enrollment into the study. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the study treatment.
* Karnofsky/Lansky performance status ≥ 50 %
* Adequate organ function as defined below:

  * Total bilirubin ≤ 2 mg/dL
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine within normal institutional limits OR creatinine clearance ≥ 50 mL/min/1.73 m2 by Cockcroft-Gault Formula (adults) or Schwartz formula (pediatric cohort)
  * Oxygen saturation ≥90% on room air
  * Ejection fraction ≥35%
* Able to be off corticosteroids and any other immune suppressive medications beginning on Day -3 and continuing until 30 days after the infusion of the CIML NK cells. However, use of low-level corticosteroids is permitted if deemed medically necessary. Low-level corticosteroid use is defined as 10mg or less of prednisone (or equivalent for other steroids) per day.
* Women of childbearing potential must have a negative pregnancy test within 28 days prior to study registration. Female and male patients (along with their female partners) must agree to use two forms of acceptable contraception, including one barrier method, during participation in the study and throughout the DLT evaluation period.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Relapsed after allogeneic transplantation.
* Isolated extramedullary relapse (phase II only).
* More than one course of salvage chemotherapy for primary induction failure or AML relapsing after CR1 (phase II only).
* Circulating blast count ≥30,000/µL by morphology or flow cytometry (cytoreductive therapies including leukapheresis or hydroxyurea are allowed).
* Uncontrolled bacterial or viral infections, or known HIV, Hepatitis B or C infection.
* Uncontrolled angina, severe uncontrolled ventricular arrhythmias, or EKG suggestive of acute ischemia or active conduction system abnormalities.
* New progressive pulmonary infiltrates on screening chest x-ray or chest CT scan that have not been evaluated with bronchoscopy. Infiltrates attributed to infection must be stable/ improving after 1 week of appropriate therapy (4 weeks for presumed or proven fungal infections).
* Known hypersensitivity to one or more of the study agents.
* Received any investigational drugs within the 14 days prior to the first dose of fludarabine.
* Pregnant and/or breastfeeding.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Cashen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper MA, Elliott JM, Keyel PA, Yang L, Carrero JA, Yokoyama WM. Cytokine-induced memory-like natural killer cells. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1915-9. doi: 10.1073/pnas.0813192106. Epub 2009 Jan 30. PMID 19181844
- [Background] Romee R, Schneider SE, Leong JW, Chase JM, Keppel CR, Sullivan RP, Cooper MA, Fehniger TA. Cytokine activation induces human memory-like NK cells. Blood. 2012 Dec 6;120(24):4751-60. doi: 10.1182/blood-2012-04-419283. Epub 2012 Sep 14. PMID 22983442
- [Background] Ni J, Miller M, Stojanovic A, Garbi N, Cerwenka A. Sustained effector function of IL-12/15/18-preactivated NK cells against established tumors. J Exp Med. 2012 Dec 17;209(13):2351-65. doi: 10.1084/jem.20120944. Epub 2012 Dec 3. PMID 23209317
- [Derived] Berrien-Elliott MM, Becker-Hapak M, Cashen AF, Jacobs M, Wong P, Foster M, McClain E, Desai S, Pence P, Cooley S, Brunstein C, Gao F, Abboud CN, Uy GL, Westervelt P, Jacoby MA, Pusic I, Stockerl-Goldstein KE, Schroeder MA, DiPersio JF, Soon-Shiong P, Miller JS, Fehniger TA. Systemic IL-15 promotes allogeneic cell rejection in patients treated with natural killer cell adoptive therapy. Blood. 2022 Feb 24;139(8):1177-1183. doi: 10.1182/blood.2021011532. PMID 34797911
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * 2 patients enrolled in the Phase I portion of the trial relapsed and were re-enrolled as compassionate use patients and are only included in the enrollment numbers once.
  * With amendment 16, the decision was made to return to the use of rhIL-2 support instead of ALT-803.
Groups:
- Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells: * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors over 5 hours on day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion over 15-60 minutes on day 0.
  * Interleukin-2: Patients receive aldesleukin SC every other day for 2 weeks starting on day 1 (total of 7 doses)
- Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells: * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors on Day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion on Day 0.
  * Subcutaneous ALT-803 will begin approximately 4 hours after the infusion and will continue for a total of 2 doses (Days 0 and 5).
- Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells: The recipient will begin a lymphodepleting preparative regimen of fludarabine and cyclophosphamide on Day -6. The haploidentical donor identified by HLA matching of the immediate family members will undergo non-mobilized large volume (20-L) leukapheresis on Day -1, and the NK cell product will be infused into the recipient on Day 0. Subcutaneous IL-2 will begin approximately 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses.
- Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells: * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors on Day -1
  * CIML NK Cells: Patients undergo CIML NK cell infusion on Day 0
  * Subcutaneous IL-2 will begin approximately 2-4 hours after infusion and will continue every other day through Day 12 for a total of 7 doses
Period: Overall Study
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells | Donors
Started | 5 | 5 | 9 | 8 | 9 | 8 | 45
Completed | 3 | 4 | 5 | 8 | 9 | 8 | 45
Not Completed | 2 | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 4 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells | Donors | Total
Number analyzed (Participants) | 5 | 5 | 9 | 8 | 9 | 8 | 45 | 89
Age, Continuous [Median (Full Range); unit: years] | 76 [70 to 77] | 72 [51 to 76] | 71 [43 to 83] | 62.5 [52 to 77] | 71 [18 to 83] | 13 [2 to 16] | 46 [25 to 70] | 52 [2 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5 | 3 | 3 | 22 | 38
  Male | 4 | 3 | 7 | 3 | 6 | 5 | 23 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 5 | 5 | 8 | 8 | 9 | 7 | 38 | 80
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 7
  White | 3 | 5 | 8 | 7 | 8 | 7 | 36 | 74
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 9 | 8 | 9 | 8 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated or Tested Dose (MT/TD) of CIML-NK Cells (Phase I)
Description: Defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity (DLT) or the maximum dose if less than or equal to 1 patient suffers a DLT at the maximum dose.
Time Frame: 35 days
Measure: Number; unit: x 10^7 cells/kg
Groups:
- Phase I: * Lymphodepleting Preparative Regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on days -5 and -4.
  * Donor Leukapheresis: Peripheral blood cells are collected from haploidentical related donors over 5 hours on day -1.
  * CIML NK Cells: Patients undergo CIML NK cell infusion over 15-60 minutes on day 0.
  * Interleukin-2: Patients receive aldesleukin SC every other day for 2 weeks starting on day 1 (total of 7 doses)
Arm/Group | Phase I
Number analyzed (Participants) | 19
x 10^7 cells/kg | 1.0

2. Primary Outcome: Complete Remission Rate (CR/CRi) in Participants With Relapsed or Refractory AML Following CIML NK Therapy (Phase II)
Description: * Complete remission rate (CR): Morphologically leukemia free state (i.e. bone marrow with <5% blasts by morphologic criteria and no blasts with Auer rods, no evidence of extramedullary leukemia) and absolute neutrophil count ≥1000 /μL and platelets ≥100,000 /μL. Patient must be independent of transfusions
  * Complete Remission with Incomplete Blood Count Recovery (CRi): All of the above criteria for CR must be met, except that absolute neutrophils <1000 /μL or platelets <100,000 /μL in the blood.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 8 | 9
Participants | 0 | 3

3. Primary Outcome: Safety of CIML NK Cells as Measured by the Number of Participants With Treatment Related Adverse Events (Pediatric Cohort)
Description: * Graded using the National Cancer (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Related indicates possibly, probably, or definitely related to study treatment.
  * Adverse events will be collected from Day 0 to Day +35; however, bone marrow suppression (ANC < 500/uL/µL) and AEs of GVHD involving the liver, skin, or GI tract will be recorded to Day 100.
Time Frame: Through Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 8
Participants
  Chills : Grade 2 | 5
  Anorexia : Grade 2 | 1
  Anorexia : Grade 3 | 1
  Alanine aminotransferase increased : Grade 1 | 3
  Alanine aminotransferase increased : Grade 3 | 1
  Aspartate aminotransferase increased : Grade 1 | 1
  Aspartate aminotransferase increased : Grade 3 | 1
  Fever : Grade 3 | 3
  Hypertension : Grade 2 | 2
  Hyperammonemia : Grade 2 | 1
  Capillary leak syndrome : Grade 2 | 2
  Hypokalemia : Grade 1 | 2
  Hypophosphatemia : Grade 4 | 1
  Hypocalcemia: Grade 1 | 1
  Hypomagnesemia: Grade 1 | 1
  Hyperkalemia: Grade 1 | 1
  Headache: Grade 1 | 1
  Headache: Grade 2 | 1
  Myalgia: Grade 1 | 1
  Arthralgia: Grade 1 | 1
  Fatigue: Grade 1 | 1
  Injection site reaction: Grade 2 | 1
  Epistaxis: Grade 3 | 3
  Hematoma: Grade 1 | 1
  Paresthesia: Grade 1 | 1
  Pain: Grade 1 | 1
  Pain: Grade 2 | 1
  Sinus tachycardia: Grade 1 | 2
  Tachypnea: Grade 1 | 1
  Vomiting: Grade 1 | 1
  Skin induration: Grade 1 | 1
  Malaise: Grade 1 | 1
  Febrile neutropenia: Grade 1 | 3
  Flushing: Grade 1 | 1
  Hypoalbuminemia: Grade 1 | 1

4. Secondary Outcome: Response Assessed According to IWG Criteria (Phase 1, Phase II, and Pediatric)
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 5 | 5 | 9 | 8 | 9 | 8
Participants
  Complete remission (CR) | 1 | 2 | 0 | 0 | 0 | 0
  Complete remission with incomplete blood count recovery (CRi) | 0 | 0 | 3 | 0 | 3 | 1
  Partial remission (PR) | 0 | 0 | 0 | 0 | 0 | 0
  Stable disease (SD) | 0 | 1 | 0 | 6 | 1 | 2
  Treatment Failure (TF) | 1 | 0 | 1 | 0 | 1 | 0
  Progressive disease (PD) | 1 | 0 | 1 | 1 | 2 | 4
  Marrow complete response (mCR) | 0 | 0 | 1 | 0 | 0 | 0
  Morphologically leukemia-free state (MLFS) | 0 | 1 | 2 | 0 | 0 | 0
  Not evaluable | 2 | 1 | 1 | 1 | 2 | 1

5. Secondary Outcome: Duration of Remission (DOR) (Phase I, Phase II, and Pediatric)
Description: DOR is defined only for patients who achieve a complete remission (CR), complete remission with incomplete blood count recovery (CRi), marrow complete response (mCR), or partial remission (PR), and is measured from the first date of attaining CR or PR until the date of disease progression or death.
Time Frame: Up to 3 years
Population: Only for patients who achieve a complete remission (CR), complete remission with incomplete blood count recovery (CRi), marrow complete response (mCR), or partial remission (PR).
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 1 | 2 | 4 | 0 | 3 | 1
days | 126.0 [126 to 126] | 22.0 [-29.0 to 73.0] | 76.5 [21.0 to 208.0] |  | 30.0 [6.0 to 35.0] | 80.0 [80.0 to 80.0]

6. Secondary Outcome: Time to Progression (Phase I, Phase II, and Pediatric)
Description: TTP is defined as the time from date of first dose of fludarabine until evidence of disease progression.
Time Frame: Up to 3 years
Population: Not evaluable: 2 patients Phase 1 Dose Level 1 (didn't receive adequate cell dose, expired before infusion). 2 patients Phase I Dose Level 2 (expired before infusion, received haplo transplant before PD). 3 patients Phase I Dose Level 3 (no bone marrow biopsy, 2-expired before PD). 2 patients Phase II IL-2 (2-no bone marrow biopsy). 1 patient Phase II ALT-803 (expired before response assessment). 2 patients Pediatric (expired before PD, poor bone marrow sample).
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 7 | 6
days | 20.0 [20.0 to 187.0] | 36.0 [34.0 to 110.0] | 46.0 [20.0 to 273.0] | 34.0 [33.0 to 35.0] | 33.0 [20.0 to 61.0] | 28.0 [20.0 to 35.0]

7. Secondary Outcome: Disease Free Survival (DFS) (Phase I, Phase II, and Pediatric)
Description: DFS is defined as the time from the day CR, mCR, or CRi is documented until disease progression or death.
Time Frame: Up to 3 years
Population: Only those patients with CR, mCR, or CRi are evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 1 | 2 | 4 | 0 | 3 | 1
days | 126.00 | 73.00 [NA to NA] — Due to the small sample size (N=2), the 95% CI is not able to be estimated. | 56.00 [21.00 to 208.00] |  | 30.00 [6.00 to 35.00] | 60.00

8. Secondary Outcome: Overall Survival (OS) (Phase I, Phase II, and Pediatric)
Description: OS is defined from the date of first dose of fludarabine on this study until death.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells | Pediatric Cohort: 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 5 | 5 | 9 | 8 | 9 | 8
days | 39.00 [4.00 to 262.00] | 142.50 [20.00 to 344.00] | 49.00 [25.00 to 396.00] | 92.00 [10.00 to 187.00] | 38.00 [24.00 to 158.00] | 147.00 [53.00 to 366.00]

9. Secondary Outcome: Toxicity as Measured by the Number of Participants With Treatment Related Adverse Events (Phase I and Phase II)
Description: * Graded using the National Cancer (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Related indicates possibly, probably, or definitely related to study treatment.
  * AEs will be collected from Day 0 to Day +35; however, bone marrow suppression (ANC < 500/uL/µL) and AEs of GVHD involving the liver, skin, or GI tract will be recorded to Day 100.
Time Frame: Through Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: 1.0 x 10^7/kg CIML NK Cells | Lead-in Cohort & Phase II (ALT-803): 1.0 x 10^7/kg CIML NK Cells | Phase II (IL-2): 1.0 x 10^7/kg CIML NK Cells
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 9
Participants
  Nausea: Grade 1 | 1 | 0 | 1 | 4 | 2
  Nausea: Grade 2 | 0 | 0 | 0 | 1 | 1
  Diarrhea: Grade 1 | 1 | 0 | 0 | 2 | 0
  Diarrhea: Grade 2 | 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase increased: Grade 1 | 1 | 0 | 0 | 2 | 1
  Alanine aminotransferase increased: Grade 1 | 2 | 0 | 0 | 0 | 1
  Proteinuria: Grade 1 | 1 | 0 | 0 | 0 | 1
  Proteinuria: Grade 2 | 0 | 0 | 0 | 1 | 1
  Blood bilirubin increased: Grade 1 | 0 | 0 | 0 | 1 | 0
  Blood bilirubin increased: Grade 2 | 1 | 0 | 0 | 0 | 0
  Alkaline phosphatase increased: Grade 1 | 1 | 0 | 0 | 0 | 0
  Sinus tachycardia: Grade 2 | 1 | 0 | 0 | 0 | 0
  Febrile neutropenia: Grade 3 | 1 | 0 | 0 | 6 | 6
  Malaise: Grade 1 | 1 | 0 | 0 | 3 | 1
  Malaise: Grade 2 | 0 | 0 | 0 | 0 | 1
  Rigors after IL-2 administration: Grade 2 | 0 | 1 | 0 | 0 | 0
  Hypoxia: Grade 2 | 0 | 0 | 1 | 3 | 1
  Dyspnea: Grade 2 | 0 | 0 | 1 | 1 | 0
  Confusion: Grade 2 | 0 | 0 | 1 | 0 | 1
  Confusion: Grade 3 | 0 | 0 | 0 | 0 | 1
  Lethargy: Grade 2 | 0 | 0 | 1 | 0 | 0
  Chills: Grade 2 | 0 | 0 | 1 | 0 | 3
  Injection site reaction: Grade 1 | 0 | 0 | 1 | 1 | 1
  Injection site reaction: Grade 2 | 0 | 0 | 0 | 4 | 0
  Rigors after CIML NK cell infusion | 0 | 0 | 1 | 0 | 0
  Alopecia: Grade 2 | 0 | 0 | 1 | 1 | 0
  Fatigue: Grade 1 | 0 | 0 | 0 | 5 | 1
  Fatigue: Grade 2 | 0 | 0 | 1 | 3 | 1
  Fatigue: Grade 3 | 0 | 0 | 0 | 0 | 3
  Anorexia: Grade 1 | 0 | 0 | 0 | 0 | 1
  Anorexia: Grade 2 | 0 | 0 | 1 | 3 | 3
  Anorexia: Grade 3 | 0 | 0 | 0 | 0 | 1
  Rigors: Grade 1 | 0 | 0 | 0 | 1 | 0
  Rigors: Grade 2 | 0 | 0 | 0 | 5 | 0
  Hypotension: Grade 1 | 0 | 0 | 0 | 1 | 2
  Hypotension: Grade 2 | 0 | 0 | 0 | 0 | 1
  Insomnia: Grade 2 | 0 | 0 | 0 | 0 | 1
  Encephalopathy: Grade 3 | 0 | 0 | 0 | 0 | 1
  Wheezing: Grade 2 | 0 | 0 | 0 | 0 | 2
  Pulmonary edema: Grade 1 | 0 | 0 | 0 | 0 | 1
  Pulmonary edema: Grade 2 | 0 | 0 | 0 | 0 | 1
  Pleural effusion: Grade 2 | 0 | 0 | 0 | 0 | 1
  Cytokine release syndrome: Grade 1 | 0 | 0 | 0 | 1 | 2
  Cytokine release syndrome: Grade 2 | 0 | 0 | 0 | 2 | 2
  Capillary leak syndrome: Grade 2 | 0 | 0 | 0 | 0 | 1
  Fever: Grade 1 | 0 | 0 | 0 | 0 | 2
  Fever: Grade 2 | 0 | 0 | 0 | 1 | 0
  Vomiting: Grade 1 | 0 | 0 | 0 | 5 | 2
  Infusion related reaction: Grade 1 | 0 | 0 | 0 | 0 | 1
  Infusion related reaction: Grade 2 | 0 | 0 | 0 | 0 | 3
  Infusion related reaction: Grade 3 | 0 | 0 | 0 | 0 | 1
  Hypertension: Grade 2 | 0 | 0 | 0 | 0 | 1
  Hypertension: Grade 3 | 0 | 0 | 0 | 5 | 2
  Neutrophil count decreased: Grade 4 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count decreased: Grade 4 | 0 | 0 | 0 | 0 | 1
  White blood cell decreased: Grade 4 | 0 | 0 | 0 | 0 | 1
  Mucositis oral: Grade 1 | 0 | 0 | 0 | 3 | 2
  Mucositis oral: Grade 2 | 0 | 0 | 0 | 1 | 0
  Headache: Grade 1 | 0 | 0 | 0 | 3 | 1
  Headache: Grade 3 | 0 | 0 | 0 | 1 | 0
  Sepsis: Grade 4 | 0 | 0 | 0 | 1 | 0
  Lung infection: Grade 3 | 0 | 0 | 0 | 4 | 0
  Platelet count decreased: Grade 1 | 0 | 0 | 0 | 4 | 0
  Platelet count decreased: Grade 4 | 0 | 0 | 0 | 1 | 0
  Pulmonary alveolar hemorrhage: Grade 2 | 0 | 0 | 0 | 1 | 0
  Rash maculo-papular: Grade 1 | 0 | 0 | 0 | 1 | 0
  Abdominal pain: Grade 1 | 0 | 0 | 0 | 1 | 0
  Hyponatremia: Grade 1 | 0 | 0 | 0 | 2 | 0
  Hyponatremia: Grade 3 | 0 | 0 | 0 | 1 | 0
  Hematuria: Grade 2 | 0 | 0 | 0 | 1 | 0
  Pruritus: Grade 1 | 0 | 0 | 0 | 1 | 0
  Creatinine increased: Grade 2 | 0 | 0 | 0 | 1 | 0
  Weight loss: Grade 1 | 0 | 0 | 0 | 2 | 0
  Bacteremia (strep mitis): Grade 3 | 0 | 0 | 0 | 1 | 0
  Hypoalbuminemia: Grade 1 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: -Adverse events were collected from Day 0 to Day +35; however, bone marrow suppression (ANC < 500/uL/µL) and adverse events of GVHD involving the liver, skin, or GI tract will be recorded to Day 100. -Phase I Dose Level 1: One subject expired prior to CIML NK cell infusion and no adverse events were collected per protocol.
Description: -Adverse events & all-cause mortality were not collected for donors. All-cause mortality for all others were collected through completion of follow-up.
Arm/Group | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells | Phase I Dose Level 3: Maximum NK Cell/Number kg | Lead-in Cohort & Phase II (ALT-803): Maximum NK Cell/Number kg | Phase II (IL-2): Maximum NK Cell/Number kg | Pediatric Cohort: Maximum NK Cell/Number kg | Donors
All-Cause Mortality (participants affected / at risk) | 5/5 | 4/5 | 8/9 | 8/8 | 9/9 | 8/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/5 | 2/9 | 4/8 | 4/9 | 0/8 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 9/9 | 8/8 | 9/9 | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells (N=5) | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells (N=5) | Phase I Dose Level 3: Maximum NK Cell/Number kg (N=9) | Lead-in Cohort & Phase II (ALT-803): Maximum NK Cell/Number kg (N=8) | Phase II (IL-2): Maximum NK Cell/Number kg (N=9) | Pediatric Cohort: Maximum NK Cell/Number kg (N=8) | Donors (N=0)
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Death due to acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 3 | 0 | NA
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Cardiopulmonary arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1: 0.5 x 10^6/kg CIML NK Cells (N=4) | Phase I Dose Level 2: 1.0 x 10^6/kg CIML NK Cells (N=5) | Phase I Dose Level 3: Maximum NK Cell/Number kg (N=9) | Lead-in Cohort & Phase II (ALT-803): Maximum NK Cell/Number kg (N=8) | Phase II (IL-2): Maximum NK Cell/Number kg (N=9) | Pediatric Cohort: Maximum NK Cell/Number kg (N=8) | Donors (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 1 | 2 | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5 | 6 | 5 | 7 | 2 | NA
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | NA
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | NA
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
NSTEMI (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | NA
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 3 | NA
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | NA
Impacted cerumen (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Double vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Retinal hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 1 | 2 | NA
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3 | 2 | NA
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 1 | 4 | 6 | 2 | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Epigastric pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | NA
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 5 | 6 | 5 | 0 | NA
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 7 | 4 | 1 | NA
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | NA
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | NA
Oral ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 6 | 5 | 2 | NA
Axilla pain/swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Body aches (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Burning at femoral area (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
CVC site tender (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Chills (General disorders) | 2 | 2 | 5 | 1 | 4 | 6 | NA
Diffuse body aches (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Edema face (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Edema limbs (General disorders) | 2 | 2 | 5 | 3 | 3 | 2 | NA
Fatigue (General disorders) | 1 | 3 | 3 | 6 | 7 | 2 | NA
Fever (General disorders) | 1 | 0 | 1 | 1 | 2 | 4 | NA
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Infusion related reaction (General disorders) | 0 | 0 | 0 | 2 | 5 | 0 | NA
Injection site reaction (General disorders) | 0 | 0 | 0 | 5 | 2 | 2 | NA
Irritability (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | NA
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Malaise (General disorders) | 2 | 1 | 0 | 2 | 3 | 1 | NA
Pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 6 | NA
Rigors (General disorders) | 0 | 0 | 4 | 6 | 0 | 0 | NA
Rigors after IL-2 administration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Gallstones (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Hyperammonemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | NA
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 3 | 4 | 0 | NA
Angioinvasive fungus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Bacteremia (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | NA
Bacteremia-Rothia mucilaginosa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Candidemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | NA
E. faecium in stool (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA
HHV-6 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Influenza AH3 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Lung infection (Infections and infestations) | 1 | 0 | 1 | 4 | 0 | 1 | NA
Oral thrush (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Rhinitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Sepsis (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 0 | NA
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | NA
Skin infection (Infections and infestations) | 0 | 2 | 3 | 0 | 0 | 0 | NA
Sphingomonas in blood (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | NA
VRE enterococcus species, stool bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Bleeding from trifusion site (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 4 | 1 | NA
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 3 | 0 | NA
Foley catheter pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Pain at bone marrow biopsy site (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Scalp hematoma post fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Subarachnoid hemorrhage post fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Tenderness at bone marrow biopsy site (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | NA
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1 | 2 | 0 | 1 | 0 | NA
Alanine aminotransferase increased (Investigations) | 3 | 2 | 4 | 1 | 3 | 5 | NA
Alkaline phosphatase increased (Investigations) | 1 | 3 | 3 | 2 | 2 | 0 | NA
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 4 | 4 | 4 | 3 | NA
Blood bilirubin increased (Investigations) | 1 | 1 | 2 | 3 | 2 | 1 | NA
Cardiac troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | NA
Creatinine increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | NA
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 3 | 1 | NA
INR increased (Investigations) | 2 | 2 | 5 | 1 | 2 | 0 | NA
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 0 | 2 | 0 | NA
Platelet count decreased (Investigations) | 2 | 2 | 3 | 1 | 0 | 0 | NA
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Weight loss (Investigations) | 0 | 1 | 3 | 6 | 1 | 0 | NA
White blood cell decreased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | NA
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 4 | 7 | 2 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 2 | NA
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 1 | NA
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | NA
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 1 | NA
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 3 | 3 | 5 | NA
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 3 | 1 | 7 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | NA
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 4 | 6 | 6 | 3 | NA
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4 | 0 | 3 | NA
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 4 | 6 | 3 | 5 | NA
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 5 | 3 | 3 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | NA
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Generalized aches and pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 2 | 0 | NA
Muscle tension left side of head (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 3 | 3 | NA
Right posterior knee knot (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Disease progression of central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Decreased motor function (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | NA
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 3 | 0 | NA
Headache (Nervous system disorders) | 0 | 1 | 2 | 3 | 3 | 3 | NA
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Sinus pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Somnolence (Nervous system disorders) | 1 | 0 | 3 | 1 | 4 | 0 | NA
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Worsening blepharospasm (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | NA
Confusion (Psychiatric disorders) | 0 | 0 | 2 | 0 | 3 | 0 | NA
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1 | 2 | 0 | NA
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 0 | NA
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1 | 1 | NA
Burning with urination (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 0 | NA
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Hematuria (Renal and urinary disorders) | 0 | 2 | 3 | 4 | 4 | 0 | NA
Proteinuria (Renal and urinary disorders) | 1 | 2 | 3 | 7 | 5 | 1 | NA
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA
Paraphimosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Penile bloody discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 3 | 2 | 1 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 2 | 2 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 3 | 0 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 3 | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 3 | 3 | 2 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 4 | 0 | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Possible aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | NA
Pulmonary alveolar hemorrhage/DAH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 4 | 1 | NA
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 2 | 0 | NA
Tachypnea-intermittent (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 0 | NA
Abrasion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 0 | 0 | NA
Blister of left great toe (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | NA
Erythema around central line (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Leukemia cutis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | NA
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3 | 2 | 1 | NA
Skin breakdown (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | NA
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | NA
Skin lesions (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | NA
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 2 | NA
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | NA
Hematoma (Vascular disorders) | 1 | 0 | 0 | 2 | 1 | 1 | NA
Hypertension (Vascular disorders) | 0 | 1 | 2 | 6 | 6 | 3 | NA
Hypotension (Vascular disorders) | 0 | 3 | 3 | 2 | 6 | 3 | NA
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Subdural hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | NA
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | NA
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT01898793/Prot_SAP_000.pdf